CLINICAL TRIAL: NCT05238233
Title: The Wearing-Off Period of Pharmacological Dilation: An Addendum to the Management of Anisocoria
Brief Title: Wearing-Off Period of Pharmacological Dilation and Anisocoria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1864081
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-01

CONDITIONS: Anisocoria
MeSH Terms: conditions — Anisocoria | interventions — Tropicamide; Pilocarpine; proxymetacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Eye Dilation and Constriction (Experimental): Participants screened for hyperopia >+1 diopter using a phoropter, have their intraocular pressures measured using a tono pen, and have their iridocorneal angle measured with a gonio lens.
  Proparacaine hydrochloride 0.5% eye drops will be used to numb the eyes before measuring intraocular pressures and prior to gonio lens.
  The following day, the participant will receive one drop of tropicamide and one drop of 1% pilocarpine in the left eye.
  If the left eye has no response to the 1% pilocarpine, or if the diameter of the pupil returned to baseline size, we will ask participants to come back to the clinic on another day to have the process repeated in the right eye.
  Interventions: Drug: Tropicamide; Drug: 1% Pilocarpine; Drug: Proparacaine Hydrochloride; Device: Tono pen AVIA; Device: VG4 Gonio; Device: Reichert phoropter

INTERVENTIONS:
Drug: Tropicamide — One drop will be given to participants
Drug: 1% Pilocarpine — One drop will be given to participants
Drug: Proparacaine Hydrochloride — One drop will be given to participants
Device: Tono pen AVIA — Participant intraocular pressures measured
Device: VG4 Gonio — Participant iridocorneal angle measured
Device: Reichert phoropter — Participant screened for hyperopia >+1 diopter

SUMMARY:
Students at the School of Medicine Greenville will be asked to participate in this study.

The aim of this study is to better understand when medical imaging is needed for patients with anisocoria (unequal pupil size).

Participation in the study includes up to 3 visits over a period of one week. Each study visit will last about 30 minutes.

At the first visit, participants will be screened for hyperopia using a phoropter, have their intraocular pressures taken using a tono-pen, and have their iridocorneal angle measured using gonioscopy at the ophthalmology clinic. Proparacaine hydrochloride 0.5% eye drops will be used to numb the eyes before measuring intraocular pressures and prior to gonio lens exam. Participants will also be asked to complete three forms.

Participants will be asked to return to the clinic on a scheduled day within one week of the screening visit to have their left eye dilated. At this visit, the diameter of the pupil will be measured using a Near card in a windowless room with a set light-level. Then, the participant will receive one drop of tropicamide in the left eye. After the drops have had time to take effect, which will be about 20-30 minutes later, the diameter of the pupil will be measured again.

Participants will then be asked to return to the clinic in 3-4 hours. At this time, the diameter of the pupil will be measured again.

The third type of eye drop used in this study is 1% pilocarpine. 1 % pilocarpine will briefly constrict the eyes. One drop of 1% pilocarpine will be administered to left eye, and the change in pupillary diameter will be measured, if any. It will take about 10-15 minutes for the 1% pilocarpine to take effect.

Participants may be required to attend 2 additional 30-minute visits on a third day depending on how their eyes respond to the drops.

This study will recruit about 10-15 participants.

ELIGIBILITY:
Inclusion Criteria:

* Student at the University of South Carolina School of Medicine Greenville
* Healthy participants
* No significant ophthalmological history

Exclusion Criteria:

* a history of angle closure glaucoma, any other type of glaucoma
* any elevated eye pressure readings
* any history of intraocular surgery or procedure.
* if the participant is found to be hyperopic to >+1 diopter, has an intraocular pressure of > 22 mm Hg in either eye, or displays an iridocorneal angle where trabecular meshwork
* known allergy to natural rubber latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eye
Groups:
- Eye Dilation and Constriction - Left Eye; Eye Dilation and Constriction - Right Eye: Participants screened for hyperopia >+1 diopter using a phoropter, have their intraocular pressures measured using a tono pen, and have their iridocorneal angle measured with a gonio lens.
  Proparacaine hydrochloride 0.5% eye drops will be used to numb the eyes before measuring intraocular pressures and prior to gonio lens.
  The following day, the participant will receive one drop of tropicamide and one drop of 1% pilocarpine in the left eye.
  If the left eye has no response to the 1% pilocarpine, or if the diameter of the pupil returned to baseline size, we will ask participants to come back to the clinic on another day to have the process repeated in the right eye.
  Tropicamide: One drop will be given to participants
  1% Pilocarpine: One drop will be given to participants
  Proparacaine Hydrochloride: One drop will be given to participants
  Tono pen AVIA: Participant intraocular pressures measured
  VG4 Gonio: Participant iridocorneal angle measured
  Reichert phoropter: Participant screened for hyperopia >+1 diopter
Period: Overall Study
Arm/Group | Eye Dilation and Constriction - Left Eye | Eye Dilation and Constriction - Right Eye
Started | 11; 11 Eye | 0; 0 Eye
Completed | 10; 10 Eye | 0; 0 Eye
Not Completed | 1; 1 Eye | 0; 0 Eye

BASELINE CHARACTERISTICS:
Groups:
- Eye Dilation and Constriction: Participants screened for hyperopia >+1 diopter using a phoropter, have their intraocular pressures measured using a tono pen, and have their iridocorneal angle measured with a gonio lens.
  Proparacaine hydrochloride 0.5% eye drops will be used to numb the eyes before measuring intraocular pressures and prior to gonio lens.
  The following day, the participant will receive one drop of tropicamide and one drop of 1% pilocarpine in the left eye.
  If the left eye has no response to the 1% pilocarpine, or if the diameter of the pupil returned to baseline size, we will ask participants to come back to the clinic on another day to have the process repeated in the right eye.
  Tropicamide: One drop will be given to participants
  1% Pilocarpine: One drop will be given to participants
  Proparacaine Hydrochloride: One drop will be given to participants
  Tono pen AVIA: Participant intraocular pressures measured
  VG4 Gonio: Participant iridocorneal angle measured
  Reichert phoropter: Participant screened for hyperopia >+1 diopter
Arm/Group | Eye Dilation and Constriction
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Constricting Response to Pilocarpine 1% in the Pharmacologically Dilated Eye
Description: Measurement of pupil diameter
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Eye Dilation and Constriction
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Eye Dilation and Constriction
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT05238233/Prot_001.pdf